CLINICAL TRIAL: NCT06140381
Title: Characterization of the Neuromuscular and Biomechanical Properties of Spastic Myopathy-affected Muscles During the Generation of Passive and Active Force: the Effect of a Management Program Based on Eccentric Exercises.
Brief Title: Strengthening in Sub-acute Stroke Survivors: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinique Du Parc de Belleville (Other)
Collaborators: Henri Mondor University Hospital (Other)
Responsible Party: Principal Investigator, Belghith Kalthoum, Principal investigator, Clinique Du Parc de Belleville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2022-A00436-37
Record Dates: First submitted 2023-11-06; First posted 2023-11-20 (Actual); Last update posted 2023-11-20 (Actual); Status verified 2023-11

CONDITIONS: Hemiparesis;Poststroke/CVA
Keywords: Rehabilitation; Skeletal muscle; Eccentric strengthening

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTG (Active Comparator): In conventional therapy, the treatment plan is determined based on medical opinion. After admission, each patient undergoes several multidisciplinary assessments aimed at objectively determining the care based on their needs. In this group, patients received only conventional rehabilitation. This will carry out in the same manner as a regular practice of the clinic. 3 sessions per week
  Interventions: Procedure: Conventional therapy
- ETG (Experimental): In the absence of a standardized eccentric isokinetic training protocol established for hemiparetic subjects on the plantar flexor muscles, the protocol designed for this study drew inspiration from the one established by Clark and Patten. (2013) and by Harris-Love et al. (2017).This protocol allows the introduction of an eccentric stimulus for individuals who are new to this type of training and progressively advances their program to include workload levels sufficiently to stimulate muscle plasticity optimally, thereby inducing skeletal muscle adaptations. 3 sessions per week
  Interventions: Procedure: Eccentric training; Procedure: Conventional therapy

INTERVENTIONS:
Procedure: Eccentric training — The eccentric program will last for 16 weeks, with a frequency of 2 sessions per week, totalling 32 sessions. At least 1 day of rest will be required between two training sessions. The participants will be placed in the similar position of the neuromuscular assessments (reference position). The Biodex System 4 dynamometer settings for the exercise sessions were also like the settings used for the assessments. The training program will be divided into two phases: a familiarization phase and a progression phase
  Arms: ETG
Procedure: Conventional therapy — 3 sessions per week of physical therapy with musculotendinous stretching and balance rehabilitation

SUMMARY:
The goal of this study is to compare between Eccentric training and conventional therapy in sub-acute stroke survivors. The primary objective of this study is to evaluate improvements in gait speed after four months of ET in comparison to conventional therapy for patients with sub-acute stroke. Secondary objectives involve assessing: i) modifications in neuromuscular parameters of PF, ii) changes in muscle stiffness within PF during passive mobilization and active force generation, and iii) modifications in architectural parameters of PF.

DETAILED DESCRIPTION:
This study will be a single-blinded, controlled, randomized design, wherein participants will be randomly assigned to one of two groups: the Conventional Therapy Group (CTG) or the Eccentric Training Group (ETG). Both groups will undergo a comprehensive series of assessments at three key time points: Ji (initial assessment), Jint (intermediate assessment), and Jf (final assessment). The study will commence with a recruitment phase, followed by a screening phase. Subsequently, there will be a 4-week period allocated for experimental testing before the intervention, and an additional 4 weeks for experimental testing after the intervention. These assessments will encompass a wide range of evaluations, including clinical health assessments, biomechanical assessments, neuromuscular evaluations, and functional assessments

ELIGIBILITY:
Inclusion Criteria:

* Subacute hemiparesis (> 3 months)
* BMI between 18.5 and 25
* Written consent to participate in the study.

Exclusion Criteria:

* Ankle impairment
* Botulinum toxin injections in PF within the last 4 months before study inclusion
* Medical contraindication for maximal effort
* Neurodegenerative disorders
* Cardiovascular disorders
* History of epilepsy.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
gait speed (m/s) through the 10-meter walking test. | initial assessment in the first week of the inclusion, intermediate assessment at 6 weeks of the inclusion, and final assessment at 12 weeks of the inclusion
  An analysis of the walking pattern will be conducted to quantify the evolution of spatio-temporal and barometric parameters of walking and their asymmetry.

SECONDARY OUTCOMES:
Biomechanical proprieties | initial assessment in the first week of the inclusion, intermediate assessment at 6 weeks of the inclusion, and final assessment at 12 weeks of the inclusion
  muscle stiffness, as expressed by the shear modulus (µ, in Kpa), will be assessed during passive ankle joint mobilization from dorsiflexion to plantar flexion and during maximal voluntary isometric contraction of Plantar flexors
Structural parameters | initial assessment in the first week of the inclusion, intermediate assessment at 6 weeks of the inclusion, and final assessment at 12 weeks of the inclusion
  Fascicle length and thickness (mm) will be assessed using the ultrasound scanner.
Neuromuscular parameters | initial assessment in the first week of the inclusion, intermediate assessment at 6 weeks of the inclusion, and final assessment at 12 weeks of the inclusion
  Peak force (N/m), submaximal force (N/m) and rate of force development (N/m) will be evaluated using the BIODEX isokinetic device during maximal volontary contraction
Functional parameters | initial assessment in the first week of the inclusion, intermediate assessment at 6 weeks of the inclusion, and final assessment at 12 weeks of the inclusion
  maximal range of motion (deg/s) , defined as the extent of stretch that the participant can comfortably endure during the stretching maneuver, will be measured using the BIODEX isokinetic device

CONTACTS AND LOCATIONS:
Overall Officials: Fedele Jean Michel, Investigator, Principal Investigator — Clinique Du Parc de Belleville
Locations (1):
- Wael Maktouf, Créteil, France

IPD SHARING:
Plan to Share IPD: No
Data will be shared upon request from researchers